CLINICAL TRIAL: NCT06905470
Title: The Effects of Eccentric Compared to Standard Strength Training in Primary Spinal Cord Injury Rehabilitation - a Matched-Pair Randomized Controlled Trial
Brief Title: The Effects of Eccentric Compared to Standard Strength Training in Primary Spinal Cord Injury Rehabilitation
Acronym: KREHA3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-21; SNCTP000006132 (Other: Swiss National Clinical Trials Portal)
Record Dates: First submitted 2025-03-05; First posted 2025-04-01 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injury
Keywords: eccentric training; strength training; upper body; aerobic performance; muscle volume
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Matched-pair randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric arm-crank (KREHA) training (Experimental): The eccentric training intervention consists of 20 training sessions performed on a symmetric arm-crank (Krafttraining mittels exzentrischer Handkurbel, KREHA) device. The training sessions have a duration of approximately 30 min and will be completed within twelve weeks, with a maximum of three sessions per week.
  Interventions: Procedure: Eccentric (KREHA) training
- Standard clinical routine strength (STAN) training (Active Comparator): The standard strength training intervention consists of a total of 20 training sessions at the gym of the study center, performed following clinical routine procedures. The training sessions have a duration of approximately 60 min and will be completed within twelve weeks, with around three sessions per week.
  Interventions: Procedure: Standard clinical routine strength (STAN) training

INTERVENTIONS:
Procedure: Eccentric (KREHA) training — 20 eccentric resistance training sessions will be performed on a symmetric arm-crank ergometer in a supine position.
  Arms: Eccentric arm-crank (KREHA) training
Procedure: Standard clinical routine strength (STAN) training — The regular strength training intervention consists of a total of 20 training sessions at the gym of the study center, performed following clinical routine procedures.
  Arms: Standard clinical routine strength (STAN) training

SUMMARY:
The goal of this clinical trial is to assess the effects of eccentric arm-crank (KREHA) training compared to standard clinical routine strength (STAN) training in individuals undergoing primary spinal cord injury (SCI) rehabilitation.

The main questions this trail aims to answer are:

* what are the effects of the training on upper body strength, aerobic performance, muscle volume, functional independence, and health-related quality of life?
* is the KREHA training feasible to implement into the rehabilitation routine?

Participants will:

* perform either 20 KREHA sessions or 20 STAN sessions within 12 weeks
* perform a test battery to collect data on training effects before (pretest) and after (posttest) the study intervention

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* informed consent as confirmed per signature.
* traumatic or disease-related SCI.
* participating in the routine strength training program during primary SCI rehabilitation at the study center (generally this is initiated around one month after SCI onset).
* wheelchair dependency during activities of daily living, defined by a score of 0-2 in the SCIM subsection regarding "Mobility in the house".
* passed sports medical assessment and having sufficient biceps/triceps function to perform arm-crank training, as determined by an experienced sports medicine physician

Exclusion Criteria:

* inflammatory or neurodegenerative diseases (including multiple sclerosis or Guillain-Barré syndrome).
* comorbidities or other health issues that may interfere with study participation, inability or contraindications to undergo the investigated intervention.
* MRI contraindications (magnetic metal parts or electronic implants such as pacemakers in the body).
* pregnancy (anamnestic).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Upper body strength | < 1 week pre and 12 weeks post intervention start.
  Change in upper body strength will be measured by a one-repetition maximum (1RM) bench press (in kg). The maximum amount of weight that can be pushed upwards for one repetition, while lying in a supine position on a weight training bench.

SECONDARY OUTCOMES:
Upper body strength | < 1 week pre and 12 weeks post intervention start.
  Change in upper body strength measured by a 1RM bench pull (in kg). The maximum amount of weight that can be pulled upwards for one repetition, while lying in a prone position on a weight training bench.
Handgrip strength | < 1 week pre and 12 weeks post intervention start.
  Change in maximum strength of three handgrip measurements (in kg) of both hands using a Jamar Handgrip Dynamometer.
Aerobic performance | < 1 week pre and 12 weeks post intervention start.
  Change in cardiopulmonary adaptations, measured by aerobic performance in an exercise test on a regular arm-crank ergometer. A ramp protocol starting at 20 Watt followed by 1 Watt / 6 sec increments to failure will be used. The following parameters will be evaluated during this aerobic endurance test: power at failure at the end of the test (in Watt), peak oxygen uptake during the test (in ml/kg/min), maximal heart rate (bpm)
Muscle volume | < 1 week pre and 12 weeks post intervention start.
  Magnetic resonance imaging (MRI) of relevant upper body muscles of the dominant upper arm and shoulder will be used to measure change in muscle volume.
Arm circumference | < 1 week pre and 12 weeks post intervention start.
  Change in arm circumference of the right and left lower and upper arm (in cm), will be used to estimate muscle volume.
Functioning during activities of daily living | < 1 week pre and 12 weeks post intervention start.
  Change in functioning during activities of daily living will be assessed by the Spinal Cord Independence Measure (SCIM) as extracted from clinical records. The SCIM total score ranges from 0-100, with higher scores indicating higher levels of functional independence.
Health-related quality of life | < 1 week pre and 12 weeks post intervention start.
  Change in health-related quality of life will be assessed using the Short Form Health Survey (SF-12). Weighted physical and mental component scores range from 0-100, with higher scores indicating better physical or mental health.

OTHER OUTCOMES:
Feasibility of the KREHA training (total number of training sessions) | Throughout the intervention phase, week 0-12
  Successful implementation of the KREHA training in the clinical routine, by assessing whether the 20 KREHA sessions are completed within 12 weeks.
Feasibility of the KREHA training progression (number of sessions adapted) | Throughout the intervention phase, week 0-12
  Feasibility of the KREHA training progression, by assessing how many training sessions needed to be adapted.
Feasibility of the KREHA training progression (power adaptation) | Throughout the intervention phase, week 0-12
  Feasibility of the KREHA training progression, by assessing how much the target power (in Watts) of a training session needed to be adapted compared to the initially planned progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No